CLINICAL TRIAL: NCT05910775
Title: Role Of Non-Specific Effects in The Treatment of Depression With Esketamine
Acronym: ROSETTE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was suspended due to challenges in recruiting a sufficient number of participants within a reasonable timeframe. Despite our efforts, enrollment did not meet the required threshold to proceed as planned.
Sponsor: Yale University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2000034829; 2UL1TR001863-06 (NIH)
Record Dates: First submitted 2023-06-06; First posted 2023-06-20 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Depressive Episode
MeSH Terms: interventions — Lead

STUDY DESIGN:
Intervention Model Description: Patients who are deemed clinically appropriate for esketamine will be approached for participation in the study.
Who Masked: Outcomes Assessor
Masking Description: Only outcome assessors collecting MADRS are masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (No Intervention): Participants receive TAU
- Intervention + TAU (Experimental): Participants receive a presentation prior to the first treatment and receive a "follow up" session within 24 hours after the first treatment in addition to treatment as usual
  Interventions: Behavioral: Pre and Post Treatment Presentations

INTERVENTIONS:
Behavioral: Pre and Post Treatment Presentations — A short presentation provided to the participants within 72 hours prior to the first treatment of the acute course. The presentation will emphasize the effectiveness of the treatment, and provide notable encouragement and reassurance. The intervention group will additionally receive a follow up session within 24 hours after the first treatment to provide encouragement and reassurance
  Arms: Intervention + TAU

SUMMARY:
The investigators aim to examine the magnitude of non-specific effects in the treatment of depressive episodes with esketamine, by providing patients in the intervention group with a pretreatment presentation and post-treatment follow up session, to assess whether nonspecific effects can be used effectively to improve the effectiveness of treatment with esketamine.

DETAILED DESCRIPTION:
Primary Objective:

To determine whether a positive presentation before first treatment improves expectation of improvement from treatment in patients receiving esketamine for a depressive episode within 24 hours after the first treatment.

Secondary Objectives:

To determine whether a post-treatment follow up session to provide encouragement and reassurance improves expectation of improvement from treatment in patients receiving esketamine for a depressive episode within 24 hours after the first treatment.

To determine whether a positive presentation results in an improved response from treatment in patients receiving esketamine for a depressive episode as measured by MADRS score within 24 hours after the first treatment.

To determine whether a positive presentation before first treatment, combined with a posttreatment follow up session after first treatment, result in an improved response from treatment in patients receiving esketamine for a depressive episode as measured by MADRS score by the end of the acute course of esketamine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be either male or female and at least 18 years old
* Deemed clinically appropriate to receive esketamine by a Yale Interventional Psychiatry physician.
* Written consent for the study procedures
* Ability and willingness, in the investigator's judgement, to comply with the study schedule, treatment plan, and other trial requirements for the duration of the study.

Exclusion Criteria:

* Hearing or visual impairment to the degree that would interfere with ability to view the presentation
* Difficulty in understanding spoken or written English
* Unable to provide informed consent
* Dementia or other cognitive disorder or intellectual disability that would impair the subject's ability to understand the presentation (per investigator judgment)
* Any other medical or psychiatric comorbidity that the investigator judges would put the participant at additional undue risk due to study participation or would impair subject's ability to participate in the study.
* Previous Esketamine or ketamine treatment
* Unable to give informed consent
* Was previously enrolled/randomized into the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-07-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sina Nikayin, MD, Principal Investigator — Yale University
Locations (1):
- Yale Psychiatry Hospital Interventional Psychiatry Services (IPS) unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Period: Overall Study
Arm/Group | Treatment as Usual (TAU) | Intervention + TAU
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual (TAU) | Intervention + TAU | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Group Difference in Change in Question 6 Score on Treatment Credibility and Expectancy Scale (CEQ-6)
Description: Participants' expectations will be assessed by the change in the group score of item 6 of the CEQ-6 at baseline and after the presentation (before treatment 1). Item 6 is scored from 0% (not at all) to 100% (very much). Higher scores indicates expectations have been met.
Time Frame: baseline and after presentation (before treatment 1), up to 30 days
Population: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Treatment as Usual (TAU) | Intervention + TAU
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Group Difference in Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Score
Description: MADRS score will be used to assess whether a positive presentation results in an improved response from treatment in participants receiving esketamine for a depressive episode within 24 hours after the first treatment. MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. Each item is rated on a 0-6 scale, resulting in a maximum total score of 60 points, with higher scores indicative of greater depressive symptomology.
Time Frame: baseline and within 24 hours post treatment 1
Population: as for baseline characteristics
Arm/Group | Treatment as Usual (TAU) | Intervention + TAU
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Treatment as Usual (TAU) | Intervention + TAU
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT05910775/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT05910775/ICF_001.pdf